CLINICAL TRIAL: NCT01525225
Title: Evaluation of the Pharmacokinetics of Saxagliptin, 5-Hydroxy Saxagliptin, and Metformin in Children and Adolescents Aged 10 to 17 Years With Type 2 Diabetes Mellitus Following Oral Administration of Saxagliptin and Metformin XR Fixed Dose Combination Tablet and Co-Administration of Saxagliptin and Glucophage® (Metformin) IR Tablets
Brief Title: Study of Saxagliptin, 5-Hydroxy Saxagliptin, and Metformin Concentrations/Levels in Pediatric Subjects With T2DM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Release of Post Marketing Requirement for this study. Terminated November 2013.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CV181-153
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC (Experimental)
  Interventions: Drug: Metformin immediate release (IR); Drug: Saxagliptin; Drug: Metformin IR; Drug: Saxagliptin/Metformin XR FDC; Drug: Metformin XR

INTERVENTIONS:
Drug: Metformin immediate release (IR) — Tablet, Oral, 1000 mg, twice daily, 1 day
  Other Names: Glucophage® IR
Drug: Saxagliptin — Tablet, Oral, 5 mg, single-dose, 1 day
Drug: Metformin IR — Tablet, Oral, 1000 mg, twice daily, 5 days
  Other Names: Glucophage® IR
Drug: Saxagliptin/Metformin XR FDC — Tablet, Oral, 2.5 mg Saxagliptin/1000 mg Metformin extended release (XR), Single-dose of 2 tablets. Fixed dose combination (FDC).
Drug: Metformin XR — Tablet, Oral, 500 mg, Single-dose of 4 tablets
  Other Names: Glucophage® XR

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of Saxagliptin, 5-hydroxy Saxagliptin, and Metformin in pediatric subjects with Type 2 diabetes mellitus (T2DM) following oral administration of Saxagliptin and Metformin XR fixed dose combination tablet and co-administration of Saxagliptin and Glucophage® (Metformin) IR tablets

DETAILED DESCRIPTION:
The primary purpose is to assess the pharmacokinetics of Saxagliptin, 5-hydroxy Saxagliptin, and Metformin in pediatric subjects aged 10 to 17 years with T2DM following oral administration of Saxagliptin and Metformin XR fixed dose combination tablet and co-administration of Saxagliptin and Glucophage® (Metformin) IR tablets

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2DM
* Male and female subjects ages 10-17
* Body weight ≥50 kg
* Glycosylated hemoglobin (HbA1c) 6.5 to 10%

Exclusion Criteria:

* Fasting plasma glucose (FPG) > 240 mg/dL at screening
* Abnormal renal function
* Active liver disease and/or significant abnormal liver function

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Osborne Research Center, Little Rock, Arkansas
  - Axis Clinical Trials, Los Angeles, California
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - The Children'S Mercy Hospital And Clinics, Kansas City, Missouri
  - Promedica Toledo Children'S Hospital, Toledo, Ohio
  - Promedica Toledo Childrens Hospital, Toledo, Ohio
  - Childrens Hospital Of Pittsburgh Of Upmc, Pittsburgh, Pennsylvania

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon approval of Kombiglyze™ XR, the Food and Drug Administration (FDA) required the conduct of this clinical pharmacology study in pediatric patients as a post-marketing requirement (PMR). Study was initiated February 2013. On 14-Nov-13, the FDA issued a letter stating release from this PMR, thus the study was terminated prior to completion.
Pre-assignment Details: A total of 4 participants were enrolled. Two participants were treated and completed the study prior to the termination of the study.
Groups:
- Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC: Each participant received one dose of a 5 mg saxagliptin tablet once a day (QD) and a 1000 mg Glucophage® immediate release (IR) tablet twice a day (BID) on Day 1. On Days 2 through 6, participants received a 1000 mg tablet of Glucophage® IR BID, and on Day 7, participants received one dose of two 2.5 mg saxagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablets. Finally, on Day 8 participants received four 500 mg Glucophage® IR tablets QD. All study drugs were administered with food.
Period: Enrollment
Arm/Group | Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC
Started | 4
Completed | 2
Not Completed | 2
Not completed — No longer met study criteria | 1
Not completed — Other | 1
Period: Treated
Arm/Group | Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC: Each participant received one dose of a 5 mg saxagliptin tablet once a day (QD) and a 1000 mg Glucophage® IR tablet twice a day (BID) on Day 1. On Days 2 through 6, participants received a 1000 mg tablet of Glucophage® IR BID, and on Day 7, participants received one dose of two 2.5 mg saxagliptin/1000 mg metformin XR FDC tablets. Finally, on Day 8 participants received four 500 mg Glucophage® IR tablets QD. All study drugs were administered with food.
Arm/Group | Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 13.0 [10.0 to 16.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | 1
  White | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) , Serious Adverse Events (SAEs), AEs Leading to Discontinuation, Death
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Day 1 up to Day 8, plus 30 days
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC
Number analyzed (Participants) | 2
participants
  AE | 2
  Treatment-Related AE | 1
  AE Leading to Discontinuation | 0
  SAE | 0
  Death | 0

2. Secondary Outcome: Number of Participants With Marked Chemistry or Hematology Laboratory Abnormalities
Description: Lower limit of normal (LLN); upper limit of normal (ULN); treatment (RX); pre-treatment (Pre-Rx); units per liter (U/L); millimoles per liter (mmol/L). Alkaline phosphatase U/L:>1.25*Pre-RX if Pre-RX >ULN or >1.25*ULN if Pre-RX <=ULN; aspartate aminotransferase U/L: >1.25*Pre-RX if Pre-RX>ULN or 1.25*ULN if Pre-RX<=ULN;alanine aminotransferase U/L: >1.25*Pre-RX if Pre-RX>ULN or 1.25*ULN if Pre-RX<=ULN;blood urea nitrogen mmol/L: >1.1*ULN if Pre-RX <=ULN or >1.2*Pre-RX if Pre-RX >ULN; total bilirubin µmol/L: >1.1*ULN if Pre-RX <=ULN or >1.25*Pre-RX if Pre-RX >ULN; creatine phosphokinase U/L: >1.5*Pre-RX if Pre-RX>ULN or >1.5*ULN if Pre-RX <= ULN. Grams per liter (g/L); cells per liter (c/L). Hemoglobin (g/L): <0.85* pre-RX; hematocrit (%): <0.85*pre-RX;erythrocytes (*10^12 c/L): <0.85*pre-RX; platelet count (*10^9 c/L): <0.85*LLN if pre-RX>=LLN, or if Pre-Tx <LLN; leukocytes (*10^9 c/L): <0.85*LLN if pre-RX <LLN,or <0.9*LLN if LLN<=Pre-RX<=ULN.
Time Frame: Day 1 to Day 8
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 8, plus 30 days.
Description: Study initiated February 2013 and was terminated November 2013. Last patient, last visit was June 2013.
Arm/Group | Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin + Saxagliptin + Saxagliptin/Metformin XR FDC (N=2)
Headache (Nervous system disorders) | 2

LIMITATIONS AND CAVEATS:
Due to the small number of participants (2), the primary endpoints, pharmacokinetic parameters, were not calculated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.